CLINICAL TRIAL: NCT06453018
Title: Positional Therapy for Childhood Obstructive Sleep Apnoea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kate Ching Ching Chan, Associate Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POSAv1.0
Record Dates: First submitted 2023-11-01; First posted 2024-06-11 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Children aged 6 to 17 years of age with positional OSA (POSA) will receive the positional therapy.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Positional therapy
  Interventions: Device: Positional device, Rematee Bumper Belt or Night Shift

INTERVENTIONS:
Device: Positional device, Rematee Bumper Belt or Night Shift — Positional device, Rematee Bumper Belt (Rematee, Blaine, Washington), or Night Shift (Advanced Brain Monitoring) on chest belt, will be used as the intervention

SUMMARY:
Obstructive sleep apnoea (OSA) in children is a prevalent sleep disorder associated with a wide spectrum of morbidities, including neurobehavioural, cardiovascular, and metabolic complications. Positional OSA (POSA) is one of the distinct clinical phenotypes in which obstructive respiratory events occur predominantly while sleeping in the supine position. As the majority of the OSA events in POSA occur in the supine position, positional therapy has become a reasonable non-invasive treatment strategy.

The primary objectives of our study are 1) To investigate the feasibility of positional therapy in children with positional OSA; 2) To investigate the efficacy of positional therapy in children with positional OSA.

Hypothesis to be tested: 1) Positional therapy is feasible in children with positional OSA.

2) Positional therapy is efficacious in children with positional OSA by improving sleep related symptoms and quality of life.

Design and subjects: A prospective case-control study. 20 children aged 6 to 17 years of age with positional OSA (POSA) will be invited to join the study.

Primary and secondary outcome measures: The changes in sleep-related symptoms, quality of life and behavioral measures between the baseline and 3 months after treatment with a positional device therapy. Adherence to the positional device.

Statistical Analysis: Continuous data will be presented as mean and standard deviation or median with the interquartile range depending on its distribution, whereas categorical data will be shown as proportions. Changes in outcome measures between the baseline and 3 months after using the positional device will be compared using Wilcoxon signed rank tests. Within-subject differences in the outcome parameters will be tested by paired t-tests, McNemar tests, and marginal homogeneity tests for continuous, dichotomous, and categorical data respectively.

Expected results: Positional therapy is practicable and efficacious in children with positional OSA by improving sleep related symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-17 years
2. Diagnosis of positional OSA on a baseline diagnostic polysomnography (PSG), defined as 1) an overall OAHI ≥ 5 events/hour (moderate-to-severe OSA), 2) a supine OAHI greater than or equal to two times of the non-supine OAHI, and 3) at least 30 minutes or 10% of total sleep time of supine sleep, and at least 30 minutes or 10% of total sleep time of non-supine sleep observed in the diagnostic PSG (9-11)
3. Informed consent from a parent or a legal guardian

Exclusion Criteria:

1. Severe OSA with an OAHI ≥ 30 events/hour that conventional treatment such as adenotonsillectomy and CPAP should be considered before positional therapy, severe disease warranting urgent referral for treatment
2. Genetic, syndromal, or metabolic disease
3. Congenital or acquired neuromuscular disease
4. Craniofacial abnormalities
5. Structural or congenital heart disease
6. Severe chronic respiratory disease that may affect the oxygen saturation or ventilation during sleep and positional therapy is regarded as not appropriate
7. Autism spectrum disorder or severe developmental delay (developmental or functional age <66% of chronological age (16) that could affect the tolerance to the positional device
8. Current treatment with positive airway pressure
9. Skeletal abnormalities or other conditions that restrict the sleeping position

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-07-03 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep related symptoms | 3 months
  Questionnaire-based assessments on sleep symptoms by Pediatric Sleep Questionnaire (PSQ): The PSQ consists of 22 items, and responses are scored as "yes" = 1, "no" = 0, and "don't know" = missing. The mean response on non-missing items is the score, which can range from 0 to 1. Higher scores on the PSQ indicate a greater likelihood of sleep-related problems. Specifically, a score greater than 0.33 (33% of questions answered positively) suggests a high risk for pediatric sleep-related breathing disorders
Daytime sleepiness assessment 1 | 3 months
  Questionnaire-based assessments on sleep symptoms by Pediatric Daytime Sleepiness Scale (PDSS): The PDSS consists of 8 questions, each scored on a 5-point Likert scale ranging from 0 to 4. Therefore, the total score can range from 0 to 32. Higher scores on the PDSS indicate greater daytime sleepiness.
Daytime sleepiness assessment 2 | 3 months
  Questionnaire-based assessments on sleep symptoms by modified Epworth Sleepiness Scale for children and adolescents (ESS-CHAD): The ESS-CHAD consists of 8 questions, each scored on a scale from 0 to 3. Therefore, the total score can range from 0 to 24. Higher scores on the ESS-CHAD indicate greater daytime sleepiness.

SECONDARY OUTCOMES:
Quality of life measure | 3 months
  Questionnaire-based assessments on quality of life measure by Obstructive Sleep Apnoea-18 questionnaire: OSA-18. is a quality of life questionnaire used to assess the impact of obstructive sleep apnea on children. It consists of 18 items, each scored on a scale from 1 to 7. Therefore, the total score can range from 18 to 126. Higher scores on the OSA-18 indicate a worse outcome, reflecting a greater negative impact on the child's quality of life due to obstructive sleep apnea. Specifically: Scores below 60 suggest a mild impact; Scores between 60 and 80 suggest a moderate impact; Scores above 80 suggest a severe impact.
Behavioural outcomes | 3 months
  Questionnaire-based assessments on behavioural outcomes using child behavior checklist CBCL. The CBCL consists of 113 items, each scored on a 3-point scale (0 = not true, 1 = somewhat or sometimes true, 2 = very true or often true). The total score can range from 0 to 226. Higher scores on the CBCL indicate more behavioral and emotional problems.
Adherence to intervention | 3 months
  Diary-based assessments on adherence or device recorded usage if using Night Shift

CONTACTS AND LOCATIONS:
Overall Officials: Kate Ching Ching Chan, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided